CLINICAL TRIAL: NCT00455494
Title: Food-Effect Bioavailability Study of AQ-13, a Candidate Antimalarial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Organization: Tulane University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K0154-2; UR3/CCU 418652; U01CI000211 (NIH)
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Malaria
Keywords: Drug-resistant malaria; Bioavailability; Food-effect study
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AQ-13

SUMMARY:
The purpose of this study is to test the safety of a 2100 mg dose of AQ-13, a new candidate antimalarial active against drug-resistant P. falciparum infection, and to determine the effect of a standard fatty meal on the absorption of the drug from the gut and its blood levels.

DETAILED DESCRIPTION:
This is a 2-stage, randomized crossover study of a 2100 mg AQ-13 dose in healthy volunteers. Fourteen healthy volunteers will be randomized to receive the drug either on an empty stomach or after a standard fatty meal under continuous monitoring in the hospital. After a washout period of 8 weeks, the volunteers will be admitted to the hospital again to receive the same dose of the drug after a fatty meal or on an empty stomach in reverse - so each volunteer will receive AQ-13 with and without a fatty meal.

Study Population:

Healthy young men and women, 21-45 years of age who are taking no chronic medications with the exception of birth control pills will be invited to participate in this food-effect bioavailability study at the Tulane-LSU General Clinical Research Center in New Orleans. Exclusion criteria include pregnancy, breast feeding, abnormal liver or kidney function tests, anemia (Hb < 12 gm per dL), chronic medications other than birth control pills, and an abnormal baseline ECG or Holter recording.

Randomization:

Allocation codes will be generated by the biostatistician in blocks, using computer software, and will be sealed in numbered, opaque envelopes. Block sizes will be determined at random and will not be known to the study personnel. The envelopes containing the randomization codes will be hand-delivered to the study pharmacist and kept in the Research Pharmacy, which is outside the GCRC.

Blinding:

The investigators and laboratory personnel performing the laboratory tests and comparing those results, electrocardiograms and Holter recordings for AQ-13 doses will be blinded to which AQ-13 doses were administered with or without a fatty meal. However, the volunteers themselves and the nursing personnel in the GCRC will know which doses were administered with and without a fatty meal. Therefore, this is a single-blinded study.

Informed Consent:

Informed consent will be obtained from each participant before screening. According to IRB guidelines, the informed consent form will be revised at yearly intervals and whenever new information on AQ-13 or its side effects becomes available.

In-patient Procedures:

On the evening of admission, pregnancy testing will be repeated and CK will be measured before drug administration the following morning. The drug administration protocol will follow the design outlined in the FDA "Guidance for Industry" for food-effect bioavailability studies (1-2). The 2100 mg AQ-13 dose will be divided into three doses of 700 mg each to be administered once a day in the morning on an empty stomach with 240 ml water after 10 hours fasting for the empty stomach arm. For the fatty meal arm, the AQ-13 dose on day 1 will be administered within 30 minutes of a standard fatty meal, prepared as described in the FDA "Guidance" and administered with 240 ml water after 10 hours of fasting. The fatty meal should be eaten within 30 minutes and the drug should be administered 30 minutes after start of the fatty meal. For both arms, water will not be allowed for 1 hour before or after the dose; and food will not be allowed for 4 hours after the dose (2). A small needle with plastic tubing and a blood thinner will be placed in the participant's arm and kept in place with paper tape to draw blood samples. The participant will then be monitored for heart rhythm, using a Holter monitor for four days beginning at the time of the first dose, and will have an electrocardiogram taken 4 hours after each dose. The purpose of the cardiac monitoring is to test whether the drug affects the QTc interval or the heart rhythm. Three 24-hr urine samples will be collected starting at the time of the first dose.

Outpatient follow up:

After the inpatient studies at the General Clinical Research Center (GCRC), participants will be asked to return to the GCRC as outpatients twice per week for 4 weeks to give (5 ml) of blood to follow the drug levels in their blood. At the 2 week follow up visit, an electrocardiogram, Holter recording, blood testing for hematology and chemistry, and visual exam will be done. At the 4 week follow up, an additional ECG and Holter recording will be obtained.

In the second stage of the study, all in-patient and out-patient follow up procedures will be the same as in the first stage, except that the study drug will be administered on an empty stomach for volunteers who took the drug after a fatty meal in the first stage and vice versa. At least an 8 week washout period must pass between participating in the two stages of the study.

References:

1. http://www.fda.gov/oc/initiatives/hiv/hivguidance.html
2. http://www.fda.gov/cder/guidance/5194fnl.pdf

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 21-45 years of age taking no chronic medications other than birth-control pills

Exclusion Criteria:

* Pregnancy,
* Breast-feeding,
* Chronic disease

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Area under the time-concentration curve
Maximal blood concentration
Adverse events

SECONDARY OUTCOMES:
Effect on heart repolarization (QTc interval change)
Clearance
Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Donald J Krogstad, MD, Principal Investigator — Tulane University Health Sciences Center
Locations (1):
- Tulane-LSU General Clinical Research Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Mzayek F, Deng H, Mather FJ, Wasilevich EC, Liu H, Hadi CM, Chansolme DH, Murphy HA, Melek BH, Tenaglia AN, Mushatt DM, Dreisbach AW, Lertora JJ, Krogstad DJ. Randomized dose-ranging controlled trial of AQ-13, a candidate antimalarial, and chloroquine in healthy volunteers. PLoS Clin Trials. 2007 Jan 5;2(1):e6. doi: 10.1371/journal.pctr.0020006. PMID 17213921